CLINICAL TRIAL: NCT02442973
Title: Handheld 3D Lumbar Spine Navigation: A Clinical Validation Study RM002
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Collaborators: Rivanna Medical, LLC (Unknown)
Responsible Party: Principal Investigator, Mohamed Tiouririne, MD, UVA Anesthesiology Faculty, University of Virginia
Other Study IDs: Rivanna Clin-002
Record Dates: First submitted 2015-05-08; First posted 2015-05-13 (Estimated); Last update posted 2022-03-10 (Actual); Status verified 2022-03

CONDITIONS: Pregnancy
MeSH Terms: interventions — Control Groups; Radionuclide Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control group (CG):: Standard practice group
  Interventions: Procedure: Control group (CG): standard practice
- Ultrasound group (UG):: SpineView3D™ anatomical "scouting" approach
  Interventions: Procedure: Ultrasound group (UG):; Device: Accuro SpineView3D™

INTERVENTIONS:
Procedure: Control group (CG): standard practice — Standard practice group
  Other Names: CG
  Groups: Control group (CG):
Procedure: Ultrasound group (UG): — SpineView3D™ anatomical "scouting" approach
  Other Names: UG
  Groups: Ultrasound group (UG):
Device: Accuro SpineView3D™ — subject will be scanned with 'Accuro SpineView3D
  Other Names: scan
  Groups: Ultrasound group (UG):

SUMMARY:
Currently, at UVA, handheld ultrasound devices (like those used to view an unborn baby) are only two dimensional. The Accuro is a three dimensional handheld ultrasound device. This device uses sound waves to create pictures of the spine in three dimensions. This may allow the physician to view the spine in more detail for procedures such as spinal anesthesia and other diagnostic procedures. Epidural analgesia is the mainstay procedure for the management of labor pain. The precise placement of a needle or catheter in proximity to landmarks of the spinal bone anatomy is required for the procedure to succeed. The current standard of care is called the 'blind approach' (i.e. without medical imaging) and involves a physician manually palpating a patient's back to locate spinal bone landmarks. The needle is then inserted with respect to the location of the landmarks and inserted until a loss-of-resistance is manually detected. This approach, while most common, has been associated with success rates as low as 68% in obese patients (2).

Alternative methods have been investigated for this problem, including ultrasound (US) guidance, which offers real-time imaging. Several studies have demonstrated ultrasound's efficacy for spinal anesthesia (1-6). However, standard US systems are engineered to image soft tissue rather than bone structures, with the consequence that bone is imaged poorly. US images are often degraded by a number of noise sources including speckle noise, reverberations and off-axis scattering, particularly when bone is present, making visualization of bone anatomy features difficult. Moreover, arranging access to ultrasound for the purpose of spinal anesthesia alone is cumbersome. Thus, the efficacy of guided spinal anesthesia and diagnostic procedures using standard ultrasound systems is limited and the benefits that it offers are heavily dependent on the user's familiarity and skill with ultrasonography (4).

Recently, new medical imaging technologies have been developed at Rivanna Medical, LLC to address the significant clinical need for technological advances that improve the placement of spinal anesthesia, epidural analgesia and other diagnostic procedures. The Accuro is a pocket-sized and battery operated ultrasound instrument that incorporates new signal processing-based technologies for enhanced bone imaging including 3D navigation of the lumbar spine. The device is a single self-contained unit consisting of an ultrasound system, ultrasound probe, and rotatable touchscreen display. The instrument enables a SpineView3D™ technology to facilitate spinal anesthesia guidance with real-time 3D navigation of the lumbar spine anatomy.

SpineView3D™ technology facilitates image interpretation of individual 2D lumbar spine scans by automating spinal bone landmark detection and depth measurements and providing a real-time assessment of scan plane orientation in 3D. SpineView3D™ makes image interpretation and measurements of the lumbar spine anatomy simple, quick, and easy. Real-time 2D scans from either SpineView3D™ or general-purpose bone presets are formed using patent-pending BoneEnhance+™ technology. The BoneEnhance+™ technology provides images of bone anatomy at greater bone-to-tissue contrast compared with conventional ultrasound image reconstructions.

ELIGIBILITY:
Inclusion Criteria:

Patients between the ages of 18 and 40 presenting for delivery and planning epidural anesthesia

* ASA-1 and ASA-2
* BMI > 30

Exclusion Criteria:

Patients with known spinal deformities allergies to ultrasound gel

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients between the ages of 18 and 40 presenting for delivery and planning epidural anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2016-02; Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Success rates: | 1 day
  defined as successful epidural administration on the first needle insertion attempt.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Tiouririne, MD, Principal Investigator — UVA Health System
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chin KJ, Perlas A, Chan V, Brown-Shreves D, Koshkin A, Vaishnav V. Ultrasound imaging facilitates spinal anesthesia in adults with difficult surface anatomic landmarks. Anesthesiology. 2011 Jul;115(1):94-101. doi: 10.1097/ALN.0b013e31821a8ad4. PMID 21572316
- [Background] Vallejo MC, Phelps AL, Singh S, Orebaugh SL, Sah N. Ultrasound decreases the failed labor epidural rate in resident trainees. Int J Obstet Anesth. 2010 Oct;19(4):373-8. doi: 10.1016/j.ijoa.2010.04.002. Epub 2010 Aug 8. PMID 20696564
- [Background] Grau T, Leipold RW, Conradi R, Martin E. Ultrasound control for presumed difficult epidural puncture. Acta Anaesthesiol Scand. 2001 Jul;45(6):766-71. doi: 10.1034/j.1399-6576.2001.045006766.x. PMID 11421838
- [Background] Grau T, Bartusseck E, Conradi R, Martin E, Motsch J. Ultrasound imaging improves learning curves in obstetric epidural anesthesia: a preliminary study. Can J Anaesth. 2003 Dec;50(10):1047-50. doi: 10.1007/BF03018371. PMID 14656785
- [Background] Chin KJ, Karmakar MK, Peng P. Ultrasonography of the adult thoracic and lumbar spine for central neuraxial blockade. Anesthesiology. 2011 Jun;114(6):1459-85. doi: 10.1097/ALN.0b013e318210f9f8. PMID 21422997
- [Background] Karmakar MK. Ultrasound for central neuroaxial blocks. Techniques in regional anesthesia and pain management 2009;13:161-70.